CLINICAL TRIAL: NCT01467141
Title: Meal-related Insulin Aspart Therapy Versus Meal-related Human Insulin Therapy in Children 2-6 Years of Age With Type 1 Diabetes Mellitus: A Multi-centre Randomised, Open-labelled, Cross-over, Safety and Efficacy Trial
Brief Title: Safety and Efficacy of Insulin Aspart in Children With Type 1 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ANA-1415
Record Dates: First submitted 2011-11-04; First posted 2011-11-08 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin Aspart; Insulin; Insulin, Isophane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IAsp (Experimental)
  Interventions: Drug: insulin aspart; Drug: isophane human insulin
- HI (Active Comparator)
  Interventions: Drug: human insulin; Drug: isophane human insulin

INTERVENTIONS:
Drug: insulin aspart — Injected s.c. (under the skin) three times a day
  Arms: IAsp
Drug: human insulin — Injected s.c. (under the skin) 30 minutes before the meals
  Arms: HI
Drug: isophane human insulin — May be administered s.c. (under the skin) in both treatment groups thrice daily

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to evaluate safety and efficacy in children with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes
* Treatment with insulin for at least 6 months prior to inclusion
* HbA1c below or equal to 11.0 %
* Currently treated with short acting, intermediate acting, long acting human insulin or analogues or a self-mix of these insulins at least 1 month prior to inclusion

Exclusion Criteria:

* The receipt of any investigational drug within one month prior to this trial
* Recurrent severe hypoglycaemia or hypoglycaemic awareness as judged by the investigator
* Total daily insulin doses at least 1.80 IU/kg
* Treatment with oral hypoglycaemic agents
* Known or suspected allergy to trial product or related products

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2002-06-19 (Actual); Primary Completion 2003-10-15 (Actual); Study Completion 2003-10-15 (Actual)

PRIMARY OUTCOMES:
Incidence of hypoglycaemic episodes during the treatment | Week 0; week 24
Change in HbA1c (glycosylated haemoglobin A1c) | Week 0; week 24

SECONDARY OUTCOMES:
Incidence of Adverse Events (AEs) | Week 0; week 24

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (6):
- Germany (6):
  - Novo Nordisk Investigational Site, Berlin
  - Novo Nordisk Investigational Site, Dresden
  - Novo Nordisk Investigational Site, Hagen
  - Novo Nordisk Investigational Site, Hamburg
  - Novo Nordisk Investigational Site, Hanover
  - Novo Nordisk Investigational Site, Osnabrück

REFERENCES:
- [Result] Danne T, Rastam J, Odendahl R, Nake A, Schimmel U, Szczepanski R, Moeller J, Deiss D. Parental preference of prandial insulin aspart compared with preprandial human insulin in a basal-bolus scheme with NPH insulin in a 12-wk crossover study of preschool children with type 1 diabetes. Pediatr Diabetes. 2007 Oct;8(5):278-85. doi: 10.1111/j.1399-5448.2007.00261.x. PMID 17850471
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com